CLINICAL TRIAL: NCT07391501
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Nitroglycerin Ointment for Postoperative Pain Relief After Endoscopic Rubber Band Ligation of Internal Hemorrhoids
Brief Title: Nitroglycerin Ointment for Pain Relief After Endoscopic Hemorrhoid Band Ligation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ying Zhu (Other)
Responsible Party: Sponsor-Investigator, Ying Zhu, Principal Investigator, Department of Internal Medicine, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYSZYYEC2026K010R001
Record Dates: First submitted 2026-01-25; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Internal Hemorrhoids; Postoperative Pain After Endoscopic Rubber Band Ligation
Keywords: Internal Hemorrhoids; Endoscopic Rubber Band Ligation; Postoperative Pain; Nitroglycerin Ointment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin Ointment Group (Experimental): Participants in this arm will receive standard perioperative management following endoscopic rubber band ligation for internal hemorrhoids, plus topical nitroglycerin ointment. The ointment will be applied to the intrarectal wound area starting after the procedure, three times daily, with approximately 1-1.5 cm of ointment per application, for a total duration of 2 weeks. Rescue analgesia with oral loxoprofen sodium will be permitted according to the predefined protocol when clinically indicated.
  Interventions: Drug: Nitroglycerin Ointment
- Placebo Ointment Group (Placebo Comparator): Participants in this arm will receive standard perioperative management following endoscopic rubber band ligation for internal hemorrhoids, plus a placebo ointment identical in appearance to the study drug. The placebo ointment will be applied to the intrarectal wound area starting after the procedure, three times daily, with approximately 1-1.5 cm of ointment per application, for a total duration of 2 weeks. Rescue analgesia with oral loxoprofen sodium will be permitted according to the predefined protocol when clinically indicated.
  Interventions: Drug: Placebo Ointment

INTERVENTIONS:
Drug: Nitroglycerin Ointment — Nitroglycerin ointment will be applied locally to the intrarectal wound area after endoscopic rubber band ligation for internal hemorrhoids. Treatment will begin immediately after the procedure. Participants will apply approximately 1-1.5 cm of ointment three times daily for a total duration of 2 weeks, in addition to standard perioperative management. Rescue analgesia with oral loxoprofen sodium will be permitted according to the predefined protocol when clinically indicated.
  Arms: Nitroglycerin Ointment Group
Drug: Placebo Ointment — A placebo ointment identical in appearance and packaging to the study drug will be applied locally to the intrarectal wound area after endoscopic rubber band ligation for internal hemorrhoids. Treatment will begin immediately after the procedure. Participants will apply approximately 1-1.5 cm of ointment three times daily for a total duration of 2 weeks, in addition to standard perioperative management. Rescue analgesia with oral loxoprofen sodium will be permitted according to the predefined protocol when clinically indicated.
  Arms: Placebo Ointment Group

SUMMARY:
This study is designed to evaluate whether nitroglycerin ointment can reduce pain after endoscopic rubber band ligation for internal hemorrhoids. Endoscopic rubber band ligation is a commonly used, minimally invasive treatment for internal hemorrhoids, but postoperative anal pain is a frequent and sometimes severe complication that can affect daily activities and recovery.

Participants undergoing endoscopic rubber band ligation will be randomly assigned to receive either nitroglycerin ointment or a placebo ointment applied locally after the procedure. Both participants and investigators will be blinded to the treatment assignment. All participants will receive the same standard perioperative care, and rescue pain medication will be provided when necessary.

The primary goal of the study is to compare the proportion of patients who require rescue pain medication within 72 hours after the procedure between the two groups. Secondary outcomes include pain intensity at multiple time points, time to complete pain relief, postoperative complications, treatment-related adverse events, and overall treatment effectiveness at 30 days. The results of this study may help identify a safe and effective option for improving pain control after endoscopic treatment of internal hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years, male or female
* Diagnosis/indication: Internal hemorrhoids grade I, II, or III scheduled for endoscopic rubber band ligation
* Consent: Able and willing to participate and provide written informed consent

Exclusion Criteria:

* Compliance/assessment: Unable to understand study endpoints or complete study records/forms
* Concomitant medications: Current use of oral nitrates or calcium channel blockers
* Allergy: Known allergy to lactulose oral solution, nitroglycerin ointment, or other study-related medications
* Pregnancy/lactation: Pregnant or breastfeeding women
* Procedure tolerance: Unable to tolerate hemorrhoid band ligation, colonoscopy, or bowel preparation
* Severe comorbidities: Severe cardiac, respiratory, neurologic, or psychiatric disorders
* Legal capacity: Lacking legal capacity for civil conduct or lacking insight/judgment to provide valid consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Use of Rescue Analgesic Medication Within 72 Hours After Procedure | 0 to 72 hours after endoscopic rubber band ligation
  The primary outcome is the proportion of participants who require rescue analgesic medication within 72 hours after endoscopic rubber band ligation for internal hemorrhoids. Rescue analgesia is defined as the use of oral loxoprofen sodium tablets at least once during the postoperative period from 0 to 72 hours. The timing, dose, frequency, and cumulative amount of rescue analgesic use will be recorded for each participant.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://rs.yiigle.com/cmaid/1339971

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT07391501/Prot_SAP_000.pdf